CLINICAL TRIAL: NCT01801761
Title: A Simplified Screening Questionnaire to Detect the Existence of Severe Obstructive Sleep Apnea in Chronic Obstructive Pulmonary Disease Patients
Brief Title: A Simplified Questionnaire to Detect OSA in COPD Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 101-3555b
Record Dates: First submitted 2012-12-28; First posted 2013-03-01 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2012-12

CONDITIONS: OSA; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- develop group: previous COPD study
- validation group: consecutive COPD patients from outpatient clinics

SUMMARY:
To detect the existence of severe obstructive sleep apnea (OSA) in chronic obstructive pulmonary disease (COPD) patients, which had higher mortality and hospitalization rate, a simplified questionnaire was developed for identifying those COPD patients with severe OSA.

DETAILED DESCRIPTION:
To detect the existence of severe obstructive sleep apnea (OSA) in chronic obstructive pulmonary disease (COPD) patients, which had higher mortality and hospitalization rate, a simplified questionnaire was developed for identifying those COPD patients with severe OSA.

With patient's BMI, neck and waist circumference, snores, witnessed apnea...

Time frame suspect to enroll 5 patients in 1 month and complete 4 patients at least we need 24 months to complete 120 patients

ELIGIBILITY:
Inclusion Criteria:

* stable COPD patients

Exclusion Criteria:

* cancer exacerbation in recent 2 months pregnancy central type sleep apnea claustrophobia chronic respiratory failure

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: develop group : previous COPD cohort study validation group : consecutive COPD patient from outpatients clinics
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The efficacy of simple questionnaire to detect severe OSA in COPD patients | since Dec 1, 2012 to Dec 1, 2014 (up to 2 years)
  The main outcome of this study : calculate the sensitivity, specificity, positive predictive value, negative predictive value, ROC curve Time frame: enroll 5 patients in 1 month and complete 4 patients at least we need 24 months to complete 120 patients PSG is standard diagnostic tool and it is no safety issue in this study

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Yu Wang, MD, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial Hospital 199 Tun-Hwa N. Rd., Taipei, Taiwan
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan